CLINICAL TRIAL: NCT01937182
Title: The Efficacy of Citalopram Treatment in Acute Stroke
Acronym: TALOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Council for Independent Research (Other); The Danish Regions Medicine Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-002253-30
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2016-12

CONDITIONS: Stroke, Ischemic
Keywords: Stroke; SSRI (Selective Serotonin Reuptake Inhibitors); Serotonin; 5-HT (5-Hydroxytryptamine); Neuroprotection; MRI (Magnetic Resonance Imaging); Platelet; CT (computerized tomography); Post Stroke Depression
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Citalopram; Selective Serotonin Reuptake Inhibitors; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective Serotonin Reuptake Inhibitors (Active Comparator): Intervention Drug: Citalopram
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Intervention Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — Citalopram 10-40 mg per day administered orally
  Other Names: Selective Serotonin Reuptake Inhibitors; SSRI; Seropram®; Cipramil®
  Arms: Selective Serotonin Reuptake Inhibitors
Drug: Placebo — 1/2-2 tablets per day with no intrinsic drug activity
  Other Names: inactive drug; inactive medicine; inactive substance
  Arms: Placebo

SUMMARY:
We wish to conduct a prospective, randomized, double blind, placebo controlled multi center study of the combined neuroprotective and antithrombotic effects of SSRI treatment after stroke.

Hypotheses:

SSRI treatment commenced in the acute phase of stroke (day 0-7) protects against new thromboembolic events and leads to better rehabilitation. 600 stroke patients will be randomized in a 1:1 ratio.

The treatment and follow up period is 6 months. During these 6 months there will be 2 clinical follow up visits, one telephone control and one visit to evaluate compliance regarding medication.

DETAILED DESCRIPTION:
Design TALOS is an investigator-initiated, national multicenter randomized- and placebo-controlled, double blind trial testing citalopram in acute ischemic stroke.

Randomization Eligible patients will be randomized 1:1 to treatment with either citalopram or placebo. Treatment allocation is double-blinded based on computer-generated algorithm via a dedicated website. Patients whose treatment is stopped within 31 days after inclusion will be replaced.

Intervention and follow-up Patients randomized to citalopram will receive oral treatment with 20 mg tablets (10 mg if age ≥65 and/or reduced liver function) for 6 months with telephone contact after 2 weeks and 3 months and follow-up visits at 1 and 6 months. If patients develop depression dosage is initially doubled, followed by an additional control to evaluate effect and, if necessary, shifted to open-label antidepressant treatment. After 6 months, treatment will either stop or switch to open-label antidepressants at the discretion of the investigator.

Substudy 120 of patients will begin treatment within 12 hours after treatment with recombinant tissue plasminogen activator. These patients will receive a standard acute magnetic resonance imaging (MRI) with additional perfusion and angio sequences. The 24-hour control scan will be done using MRI instead of conventional CT.

Data monitoring When 300 patients have been included in the trial, an interim analysis will be performed. The unblinded results of this analysis will be reviewed by an independent data monitoring committee.

ELIGIBILITY:
Inclusion Criteria:

* First ever ischemic stroke
* Age 18 years or above

Exclusion Criteria:

* Hemorrhagic stroke
* Dementia or other neurodegenerative disease
* Antidepressant medical treatment within 6 months of admission
* Acute need for antidepressant treatment
* Drug abuse or other conditions that may indicate noncompliant behavior
* Liver failure (increased liver enzyme levels up to or more than 2 times upper limit)
* Renal failure (eGFR below 30 ml/min per 1.73m2)
* Hyponatremia (S-potassium below 130 mmol/l)
* Actively bleeding ulcer
* Fatal stroke or other severe co-morbidity that markedly decreases expected life span
* Prolonged corrected QT-interval (QTc above 480 ms)
* Ongoing treatment with drugs known to prolong the QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Vascular death, Transient Ischemic Attack (TIA)/stroke and myocardial infarction (combined) | 6 months
  Myocardial Infarction: STEMI (ST segment elevation myocardial infarction) and NSTEMI (non-ST segment elevation myocardial infarction)
Functional status at 6-months | 6 months
  Functional status at 6-months, measured by the modified Rankin Scale

SECONDARY OUTCOMES:
Vascular death | 6 months
Death of any cause | 6 months
TIA/stroke | 6 months
Bleeding | 6 months
  Using the Global Utilization Of Streptokinase And Tpa For Occluded Arteries definition for bleeding (GUSTO)
Myocardial infarction | 6 months
  STEMI (ST segment elevation myocardial infarction) and NSTEMI (non-ST segment elevation myocardial infarction)
Disability/dependence | 6 months
  Using the modified Rankin Scale and the Barthel Index (BI)
Physical activity | 6 months
  Using the Physical Activity Scale for the Elderly (PASE)
Cognitive and organic cerebral impairment | 6 months
  Using the Mini-Mental State Examination and the Symbol Digit Modalities Test
Fatigue | 6 months
  Using the Multidimensional Fatigue Inventory
Post-stroke depression | 6 months
  Using the Major Depression Inventory test (MDI), Global depression scale (self and clinician and Hamilton Depression Scale - 6 item (HAM-D6)
Pathological Crying | 6 months
  Using the Pathological Crying Scale
Lesion size | 6 months
  Using FLAIR positive lesion size on MRI 24 hours after treatment with Alteplase

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Andersen, DSMc, Study Chair — Aarhus University Hospital; Kristian L Kraglund, M.D., Study Director — Aarhus University Hospital; Boris Modrau, M.D., Principal Investigator — Aalborg University Hospital; Helle Iversen, DSMc, Principal Investigator — Glostrup University Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Department of Neurology, Aalborg
  - Aarhus University Hospital, Department of Neurology, Aarhus
  - Glostrup University Hospital, Department of Neurology, Glostrup Municipality

REFERENCES:
- [Background] Siepmann T, Penzlin AI, Kepplinger J, Illigens BM, Weidner K, Reichmann H, Barlinn K. Selective serotonin reuptake inhibitors to improve outcome in acute ischemic stroke: possible mechanisms and clinical evidence. Brain Behav. 2015 Sep 23;5(10):e00373. doi: 10.1002/brb3.373. eCollection 2015 Oct. PMID 26516608
- [Background] Bonaventura A, Liberale L, Vecchie A, Casula M, Carbone F, Dallegri F, Montecucco F. Update on Inflammatory Biomarkers and Treatments in Ischemic Stroke. Int J Mol Sci. 2016 Nov 25;17(12):1967. doi: 10.3390/ijms17121967. PMID 27898011
- [Background] Mortensen JK, Johnsen SP, Larsson H, Andersen G. Early Antidepressant Treatment and All-Cause 30-Day Mortality in Patients with Ischemic Stroke. Cerebrovasc Dis. 2015;40(1-2):81-90. doi: 10.1159/000435819. Epub 2015 Jul 11. PMID 26184925
- [Background] Adelborg K, Sundboll J, Videbech P, Grove EL. The Risk of Thromboembolism in Users of Antidepressants and Antipsychotics. Adv Exp Med Biol. 2017;906:351-361. doi: 10.1007/5584_2016_125. PMID 27638627
- [Derived] Vestergaard SB, Damsbo AG, Blauenfeldt RA, Johnsen SP, Andersen G, Mortensen JK. Impact of prestroke physical activity and citalopram treatment on poststroke depressive symptoms: a secondary analysis of data from the TALOS randomised controlled trial in Denmark. BMJ Open. 2023 Mar 30;13(3):e070822. doi: 10.1136/bmjopen-2022-070822. PMID 36997260
- [Derived] Kraglund KL, Mortensen JK, Damsbo AG, Modrau B, Simonsen SA, Iversen HK, Madsen M, Grove EL, Johnsen SP, Andersen G. Neuroregeneration and Vascular Protection by Citalopram in Acute Ischemic Stroke (TALOS). Stroke. 2018 Nov;49(11):2568-2576. doi: 10.1161/STROKEAHA.117.020067. PMID 30355209
- See also: Researchgate — https://www.researchgate.net/project/The-Efficacy-of-Citalopram-Treatment-in-Acute-Stroke-TALOS